CLINICAL TRIAL: NCT02206633
Title: The Validity of Ultrasound Velocity to Assess Hydration Status of Elderly Residing in Assisted Living Facilities
Brief Title: Hydration Monitor Validation in Elderly
Status: Completed | Type: Observational
Sponsor: Artann Laboratories (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH); Appalachian State University (Other)
Responsible Party: Sponsor
Other Study IDs: HME-02; 2R44AG042990 (NIH)
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2014-11

CONDITIONS: Dehydration
Keywords: dehydration
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elderly, assisted living residents: Hydration Monitor ultrasound measurements
  Interventions: Device: Hydration Monitor

INTERVENTIONS:
Device: Hydration Monitor — Measurement of the ultrasound velocity with the Hydration Monitor for specific anatomic locations. Triplicate measurements will be made for each time-point. All subjects will also be measured for bioelectrical impedance analysis (BIA) and estimation of total body water using a leg-to-leg BIA machine.

SUMMARY:
The study will aim to determine normal daily variation of the individual hydration level in longitudinal study on elderly in assisted living facility and assess a range of variation of individual hydration baselines for elderly in a normal physiologically hydrated state.

DETAILED DESCRIPTION:
The subject pool will be comprised of 100 elderly (over 65 years old), male and female subjects who are residing in assisted living center. All subjects will provide written informed consent before participation. For the day prior testing and all testing days subjects will be encouraged to follow standard hydration guidelines for older adults by consuming 1200-2400 ml/day depending upon the body weight of subjects. The application of the HM will follow specific protocol based on the prototype HM user manual for specific anatomic locations. Triplicate measurements will be made for each time-point. All subjects will also be measured for bioelectrical impedance analysis (BIA) and estimation of total body water using a leg-to-leg BIA machine. To examine within-day and between-day variability and reliability of the HM a subgroup (N=25) of the 100 initial subjects will be selected. Within-day reliability will be evaluated by taking multiple measurements (3) during the day. Between-day reliability will include measurements (same time) for three consecutive days for the subgroup of 25 subjects. BIA measures will also be included during each of the time points for both within-day and between-day.

ELIGIBILITY:
Inclusion Criteria:

* elderly ( above 65 years old)
* male and female subjects who is residing in assisted living centers

Exclusion Criteria:

* Open wounds or rashes on calf testing area
* Visibly detectable edema
* Active skin infection
* Subjects will be excluded from the study if they can't physically stand on both feet without assistance

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The subject pool will be comprised of 100 elderly (over 65 years old), male and female subjects who are residing in assisted living center
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
To observe statistically significant changes in ultrasound velocity associated with normal daily variation of the individual hydration level of elderly | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Armen Sarvazyan, PhD, Principal Investigator — CSO, Artann Laboratories
Locations (1):
- Appalachian State University, Boone, North Carolina, United States